CLINICAL TRIAL: NCT04694521
Title: Outcomes of Side-to-end Versus End-to-end Colorectal Anastomosis in Non-emergent Sigmoid and Rectal Cancers: Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour of general and laparoscopic surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zagazig university 2
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antegrade colorectal single stapler anastomosis (Experimental): open Side to end antegrade colorectal anastomosis colo rectal cancers.
  Interventions: Procedure: openSide to end colorectal anastomosis .
- open end to end colorectal stapler anastomosis (Experimental): open end to end colorectal single anastomosis in non-emergent colo rectal cancers.
  Interventions: Procedure: open end end to end stapler anastomosis

INTERVENTIONS:
Procedure: openSide to end colorectal anastomosis . — open Side to end colorectal anastomosis
  Arms: antegrade colorectal single stapler anastomosis
Procedure: open end end to end stapler anastomosis — open end to end stapler anastomosis
  Arms: open end to end colorectal stapler anastomosis

SUMMARY:
Introduction: Cancer rectum and sigmoid is increasing nowadays. Resection and anastomosis is done laparoscopic approach with various techniques of anastomosis.

Aim of this study: to compare between open side to end colorectal anastomosis versus laparoscopic end to end colorectal anastomosis in Non-emergent colo- rectal Cancers in adults as regard anastomotic leak, intestinal function and quality of life.

Patients and Methods: Randomized controlled trial was performed on patients with Non-emergent colo rectal cancers between September 2016 and September 2018.

DETAILED DESCRIPTION:
ICancer rectum prevalence comes next to bronchogenic and prostatic malignant neoplasms in male, but it is the second cancer in female following cancer breast. [1] despite the fact that 1,000,000 patients notably every year and mortality by thousands, yet patients that live from this cancer is surging in the last years due to both sumptuous appliance of investigation and novel intervention techniques. Over two thirds of rectal cancer patients survived 5 years. [2].

Colorectal surgery principles target to merge the fulfillment of well-balanced free margin resection with bowel, urinary and potency activities. [3]. Laparoscopic rectal surgery for cancer had a famed corner in recent surgery that besieged open approach [4]. Rectal surgery has many troubles. The most troubled complication is anastomotic leakage. The prevalence of anastomotic leakage following rectal resection and anastomosis may wave to 15% of cases with high morbidity and mortality [5].The inauguration of the stapler in rectal surgery assisted the anastomosis to be in a homogeneous design, decrease strain on the suture, speedy surgery, no intra-abdominal contamination, no intrusion of anastomotic site perfusion and narrow the prevalence of anastomotic leakage. [6]. Resection of rectum is linked to low anterior resection syndrome (LARS) that usually affects quality of life [7].

2. Aim of the work, gap statement and strength of the study: During rectal cancer surgery, no conclusive path of resection and anastomosis and usually followed by the surgeons according to their experience. In the current study, we have organized a randomized clinical trial to analyze the outcomes in two groups of patients with colo rectum cancers with two different laparoscopic approaches for resection and anastomosis. The primary aim was to correlate the prevalence of anastomotic leak after both interventions. The secondary aim was to appraise intestinal functional outcome and quality of life between both groups.

Patients & Methods:

3.1 Study design and study power: This is a prospective randomized controlled trial managed in the colorectal surgical units of our University Hospitals (solitary-center) between September 2016 to September 2018. A total of 74 patients diagnosed as colorectal cancer underwent openrectal cancer surgery. The patients were randomly labeled into two groups: Group (A): included 37 patients: open side to end colorectal anastomosis (SEA) and Group (B): included 37 patients: openend to end colorectal anastomosis (EEA). As percentage of leakage from previous paper [8] was 29% VS 5.4% so sample will be 37 in each group with power 80% and confidence level 95% would be suitable to reach statistical significance (p<0.05). It is a simple random sample with a balance. Patients were randomly allocated using a random sequence computer. Patients were randomly numbered in closed envelopes, which were opened just before accomplishing the anastomosis intraoperative. Patients were unaware to the any group until after the study. It is the role of registration office.

ELIGIBILITY:
Inclusion Criteria:

* 1. colo rectum adenocarcinoma proved by biopsy and histo-pathological examination.

  2. Only resections performed with immediate anastomosis, not under cover of stoma.

  3. Expected R0 resection. 4. patients >18 years ,both sex 6. No previous history of stool or flatus incontinence, and clinically normal function of anal sphincter.

Exclusion Criteria:

1. Patients younger than 18 years , Pregnant female.
2. Inability to understand the informed consent or refuse to participate or psychiatric patients.
3. Patients with recurrent cancer, Irresectable tumour, widespread loco-regional, distant metastasis ,Combination operation and Complicated cancer e.g. obstructed or perforated.
4. Cases covered by proximal stoma.
5. Patients with lesion <3 cm from anal verge or cancer involving anal sphincter
6. preoperative chemo radiotherapy
7. Previous left sided colorectal surgery or anorectal surgeries.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
: the incidence of the anastomotic leak during hospital admission and during 30 days postoperative. | 30 days
  : the incidence of the anastomotic leak during hospital admission and during 30 days postoperative.
intestinal function | 24 months after surgery.
  intestinal function and LAR score

SECONDARY OUTCOMES:
the overall postoperative morbidities | within 90 days
  the overall postoperative morbidities by clavien-dindo classification

IPD SHARING:
Plan to Share IPD: No